CLINICAL TRIAL: NCT00001351
Title: Evaluation and Long-Term Follow-Up of Patients With Acute or Chronic Inflammatory Disorders
Brief Title: Evaluation and Long-Term Follow-up of Patients With Inflammatory Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930086; 93-I-0086
Record Dates: First submitted 2006-07-12; First posted 1999-11-04 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12-15

CONDITIONS: Inflammation
Keywords: Human; Disease; Infection; Immunology; Natural History
MeSH Terms: conditions — Inflammation; Disease; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate family members of patients: immediate family members of patients with inflammatory conditions may be evaluated under this protocol
- Patients: Inflammatory conditions associated with, but not limited, to acute and chronic infections or presumed infections, and congenital or acquired immunologic disorders

SUMMARY:
This study will investigate inflammatory diseases and disorders. Inflammation is the body s immune response to many things, including infections and other acute or chronic irritants. It may also be a sign of abnormal immune function. This study will allow evaluation and long-term follow-up of such disorders to:

* Establish and maintain a group of patients that may be eligible for other NIAID protocols.
* Provide clinical training and experience for NIAID fellows.
* Provide a mechanism for NIAID staff to maintain their clinical skills.
* Serve as a starting point for new investigations of syndromes not currently under study.

Patients between 1 and 80 years of age with acute or chronic inflammation, including but not limited to viral, fungal or bacterial infections, or abnormal immune responses may be eligible for this study. Immediate family members of patients may also be enrolled for preliminary examination to see if they are affected in any way that may warrant further investigation.

All patients and family members will have a history, physical examination and laboratory tests. Depending on the results, family members may require additional tests. Patients will have additional diagnostic tests indicated for their specific disease, according to accepted medical standards. These may include routine blood and urine tests, X-rays or other imaging studies, body fluid or tissue cultures, skin tests for allergic or immune responses, and others as needed.

Treatments will include only medications approved by the Food and Drug Administration according to accepted dose schedules and delivery methods.

Patients may be requested to donate extra blood for research studies. No more than 450 cc (30 tablespoons) will be drawn from adults within a 6-week period, and no more that 7 cc (1/2 tablespoon) from children under 18 years of age in the same time period.

DETAILED DESCRIPTION:
Inflammatory disorders, including but not limited to those caused by viral, bacterial, fungal, and parasitic infections, and those associated with aberrant immunologic responses are exceedingly common acute and chronic disorders affecting humans. The pathogeneses of these various disorders are being investigated under a number of NIAID clinical research protocols. This protocol is an evaluation and long-term follow-up protocol of such disorders for the purposes of maintaining a group of patients on which LCIM investigators draw for our other various protocols. Also, this protocol may serve as a start point to studies of syndromes or diseases not being addressed by specific protocols, and therefore, can be used to evaluate family members of patients with inflammatory conditions when appropriate in order to try to understand further the disease before embarking in a specific protocol. It is anticipated that the patients will receive a degree of clinical evaluation, care and monitoring more extensive that that generally available and that specimens collected from them can sometimes be used for laboratory studies related to inflammatory conditions.

ELIGIBILITY:
* INCLUSION CRITIERIA:
* Males and females ages 2 years and older.
* Inflammatory conditions associated with, but not limited, to acute and chronic infections or presumed infections, and congenital or acquired immunologic disorders, as determined by the principal or associated investigators.
* A NIAID/LCIM investigator has an interest in the patient s illness and is willing to serve as attending physician to supervise the patient's medical care at the NIH.
* If appropriate, immediate family members of patients with inflammatory conditions may be evaluated under this protocol to determine if they may also be affected by their relative s disease.
* Willingness to participate in clinical protocols when appropriate.
* Subjects must maintain a primary physician outside NIH for non-protocol related medical complaints and for emergency medical treatment required for these or other of their disorders.
* Willingness to have samples stored and to provide tissue samples for studying immune dysregulation and for genetic analysis.
* Ablility to provide informed consent or, for the patient cohort, has a designated legally authorized representative (LAR).
* For females, not pregnant.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Inflammatory conditions associated with, but not limited, to acute and chronic infections or presumed infections, and congenital or acquired immunologic disorders@@@- If appropriate, immediate family members of patients with inflammatory conditions may be evaluated under this protocol, as a preamble to see if further investigation is warranted, what would be done under a specific protocol.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 1993-06-01 (Actual)

PRIMARY OUTCOMES:
screening of patients for other protocols | ongoing through the study
  screening of patients for other protocols,
evaluation and follow-up of interesting patients, who do not fit in our other protocols | ongoing through the study
  evaluation and follow-up of interesting patients, who do not fit in our other protocols

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1993-I-0086.html